CLINICAL TRIAL: NCT05336617
Title: Quality of Colonoscopies Under Kalinox During the COVID 19 Epidemic
Brief Title: It is Possible to Maintain the Performance of Screening Colonoscopies Under MEOPA During the Covid 19 Epidemic Period When Access to the Operating Room is Limited
Acronym: KALINOX19
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0018
Record Dates: First submitted 2022-04-19; First posted 2022-04-20 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer
Keywords: Type of anesthesia; Colonoscopy and polypectomy; Colorectal cancer; Colonoscopy quality indicator; COVID 19
MeSH Terms: conditions — Colorectal Neoplasms; COVID-19 | interventions — Colonoscopy; Meopa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: colonoscopy — A colonoscopy is an exam used to examine the colon and rectum. During a colonoscopy, a long, flexible tube is inserted into the rectum. A tiny video camera at the tip of the tube allows the doctor to view the inside of the entire colon.
  Other Names: MEOPA

SUMMARY:
Feedback: during the COVID-19 epidemic, access to operating theaters was restricted so that anesthetists and nurse anesthetists could reinforce the resuscitation workforce.

The MEOPA was used as an alternative to sedation, allowing colonoscopies to be carried out, colon polyps and colorectal cancers to be detected.

DETAILED DESCRIPTION:
Colonoscopy is a major procedure for screening for cancers and diagnosing colorectal lesions. In France, general anesthesia remains the most widely used sedation method for colonoscopy. Faced with several constraints such as difficulty of access to the operating room, length of hospitalization and contraindications to general anesthesia, several sedation methods have been adopted.

The best known is sedation by MEOPA (equimolar mixture of oxygen protoxide of nitrogen) marketed under the name of Kalinox. It is offered as a second-line treatment after general anesthesia.

Since March 2020, the COVID-19 health crisis has forced us to change our care. Faced with restricted access to the operating room (anesthetists and nurse anesthetists requisitioned to participate in the care of patients in intensive care), colonoscopy under MEOPA was offered to patients who could have benefited from general anesthesia before the crisis. This monocentric retrospective descriptive study at the CHSF (Centre Hospitalier Sud Francilien) will make it possible to assess the quality of colonoscopies performed under MEOPA in the first line.

This is a feedback, the MEOPA having allowed us to continue and maintain the performance of screening colonoscopies during the COVID 19 epidemic.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who had a colonoscopy under MEOPA between January 2019 and May 2021 at the CHSF.

Exclusion Criteria:

* Colonoscopy under general anesthesia
* Refusal of data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults patients who underwent a colonoscopy under Kalinox in the Centre Hospitalier Sud Francilien from 01/01/2019 to 05/31/2021.
Sampling Method: Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
percentage of complete colonoscopies | at day 0
  percentage

SECONDARY OUTCOMES:
Adenoma detection rate. | at day 0
  percentage
Polyp detection rate. | at day 0
  percentage
Colorectal cancer detection rate | at day 0
  percentage
Quality of colonic preparation (Boston score) | at day 0
  Breakdown into 3 groups: good (Boston Bowel Preparation SCALE 7, 8, 9), bad (Boston Bowel Preparation SCALE 4, 5, 6) and unsatisfactory (Boston Bowel Preparation SCALE 1, 2, 3)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No